CLINICAL TRIAL: NCT01571050
Title: Systemic Fluoride Bioavailability From Toothpastes Containing Calcium Carbonate or Silica as Abrasives
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Livia Maria Andaló Tenuta, Assistant Professor, Biochemistry and Cariology, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FOPFBioavailability2011
Record Dates: First submitted 2012-03-30; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Dental Fluorosis
Keywords: toothpastes; dental fluorosis; fluoride; bioavailability
MeSH Terms: conditions — Fluorosis, Dental

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Fresh NaF/SiO2 toothpaste (Experimental)
  Interventions: Drug: Fresh NaF/SiO2 toothpaste
- Purified water (Placebo Comparator)
  Interventions: Drug: Purified water
- Aged NaF/SiO2 toothpaste (Experimental)
  Interventions: Drug: Aged NaF/SiO2 toothpaste
- Fresh MFP/CaCO3 toothpaste (Experimental)
  Interventions: Drug: Fresh MFP/CaCO3 toothpaste
- Aged MFP/CaCO3 toothpaste (Experimental)
  Interventions: Drug: Aged MFP/CaCO3 toothpaste

INTERVENTIONS:
Drug: Purified water — Ingestion of 30 mL of purified water
  Arms: Purified water
Drug: Fresh MFP/CaCO3 toothpaste — Ingestion of 31.9 mg of a fresh toothpaste containing 1450 ppm total fluoride per kg body weight, diluted in 30 mL of purified water, to provide a total intake of 49.5 ug of fluoride/kg body weight.
  Arms: Fresh MFP/CaCO3 toothpaste
Drug: Fresh NaF/SiO2 toothpaste — Ingestion of 49.5 mg of a fresh toothpaste containing 1100 ppm total fluoride per kg body weight, diluted in 30 mL of purified water, to provide a total intake of 49.5 ug of fluoride/kg body weight.
  Arms: Fresh NaF/SiO2 toothpaste
Drug: Aged NaF/SiO2 toothpaste — Ingestion of 49.5 mg of a toothpaste containing 1100 ppm total fluoride per kg body weight, diluted in 30 mL of purified water, to provide a total intake of 49.5 ug of fluoride/kg body weight. The toothpaste had been previously aged to simulate one year storage at room temperature.
  Arms: Aged NaF/SiO2 toothpaste
Drug: Aged MFP/CaCO3 toothpaste — Ingestion of 31.9 mg of a toothpaste containing 1450 ppm total fluoride per kg body weight, diluted in 30 mL of purified water, to provide a total intake of 49.5 ug of fluoride/kg body weight. The toothpaste had been previously aged to simulate one year storage at room temperature.
  Arms: Aged MFP/CaCO3 toothpaste

SUMMARY:
The risk of dental fluorosis development is related to the systemic exposure to fluoride during enamel formation. Currently, diet and fluoride toothpastes are the main sources of fluoride to children at the age-risk for fluorosis development. However, when estimating the risk of fluorosis from toothpaste inadvertently ingested, it has not been considered the systemic fluoride bioavailability. Since some toothpaste formulations may contain part of fluoride as insoluble salts, the hypothesis behind this study is that only soluble fluoride in toothpastes would be absorbed when they are inadvertently ingested. To test that, adult volunteers will ingest a standardized dose of total fluoride from commercially available toothpastes, which present different concentrations of soluble fluoride. Fluoride systemic bioavailability will be assessed by the release of fluoride in saliva up to 3 hours after ingestion (as an indicator of blood fluoride) and by urinary fluoride excretion.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Good oral health
* Normal salivary flow rate

Exclusion Criteria:

* Gastric disorders
* Renal disorders

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve of salivary fluoride concentration versus time after toothpaste ingestion | 3 hours
  Saliva will be collected before and up to 3 hours after ingestion of the toothpastes or negative control. Collections (during 3 min) will be made at 0 (immediately before ingestion), 15, 30, 45, 60, 120 and 180 min after ingestion.

SECONDARY OUTCOMES:
Maximum concentration of fluoride in saliva after toothpaste ingestion | 3 hours
  Saliva collected up to 3 hours after the ingestion of toothpastes or negative control will be analyzed for fluoride concentration and the maximum concentration during this period will be recorded.
Urinary fluoride excretion (24-h) after toothpaste ingestion | 48 hours
  Urine will be collected for the 24 hours preceeding the ingestion of the toothpastes or negative control and for the 24 hours after the ingestion. The difference in the amount of fluoride excreted in 24h urine samples, after or before the treatments, will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Livia MA Tenuta, PhD, Principal Investigator — Piracicaba Dental School, University of Campinas
Locations (1):
- Piracicaba Dental School, University of Campinas, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Background] Cury JA, Del Fiol FS, Tenuta LM, Rosalen PL. Low-fluoride dentifrice and gastrointestinal fluoride absorption after meals. J Dent Res. 2005 Dec;84(12):1133-7. doi: 10.1177/154405910508401208. PMID 16304442
- [Background] Cury JA, Oliveira MJ, Martins CC, Tenuta LM, Paiva SM. Available fluoride in toothpastes used by Brazilian children. Braz Dent J. 2010;21(5):396-400. doi: 10.1590/s0103-64402010000500003. PMID 21180793
- [Background] Martins CC, Oliveira MJ, Pordeus IA, Cury JA, Paiva SM. Association between socioeconomic factors and the choice of dentifrice and fluoride intake by children. Int J Environ Res Public Health. 2011 Nov;8(11):4284-99. doi: 10.3390/ijerph8114284. Epub 2011 Nov 10. PMID 22163207
- [Derived] Falcao A, Tenuta LM, Cury JA. Fluoride gastrointestinal absorption from Na2FPO3/CaCO3- and NaF/SiO2-based toothpastes. Caries Res. 2013;47(3):226-33. doi: 10.1159/000346006. Epub 2012 Dec 29. PMID 23295625